CLINICAL TRIAL: NCT04188951
Title: HFHS-1801-A Pilot Study of Immunotherapy As Consolidation Therapy for Patients with Recurrent Head and Neck Cancer High Risk Pathologic Features Following Surgical Salvage and Are Not Eligible for Post-operative Radiation Therapy
Brief Title: HFHS-1801-A Pilot Study of Immunotherapy As Consolidation Therapy for Patients with Recurrent Head and Neck Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Haythem Ali, M.D., Principle Investigator, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFHS-1801
Record Dates: First submitted 2019-10-31; First posted 2019-12-06 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Neoplasms
Keywords: Recurrent Head and Neck Cancer; Recurrent Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab 25 MG/1 ML Intravenous Solution [KEYTRUDA] (Other)
  Interventions: Drug: Pembrolizumab 25 MG/1 ML Intravenous Solution [KEYTRUDA]

INTERVENTIONS:
Drug: Pembrolizumab 25 MG/1 ML Intravenous Solution [KEYTRUDA] — Patients will receive 17 cycles of pembrolizumab via IV infusion of 200 mg over a period of 30 minutes, every 3 weeks starting no later than 90 days from the date of salvage head and neck therapy.

SUMMARY:
The study is a pilot study to explore the feasibility and efficacy of immunotherapy following salvage surgery for recurrent head and neck cancer.

DETAILED DESCRIPTION:
Approximately 30-40% of patients treated with a curative intent for locally advanced squamous cell carcinoma of the head and neck cancer will experience an isolated loco-regional recurrence or a second primary tumor in the previously radiated tissues1-5. Patients with recurrent head and neck cancer frequently recur locally and are still amenable for curative interventions. The current recommendations for treatment of these recurrent and second primary tumors includes surgical resection whenever possible as this has been shown to have a significantly better outcome as compared to patients treated non-surgically with radiation therapy with or without concurrent chemotherapy.

Immunotherapy is expected to be more effective with smaller amounts of disease and application of therapy when disease burden is minimal is expected to yield improved outcomes. Many trials underway at the present time explore the use of immunotherapy in earlier stages of head and neck cancer than the ones already studied. However, patients undergoing salvage therapy are understudied and no major cooperative group or industry trial is addressing this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older, of either gender, with the ability to consent to participation in the study.
* Patients must have a history of squamous cell carcinoma of the head and neck involving any sub-site in the head and neck area except nasopharynx, paranasal sinuses, and salivary gland tumors.
* All patients must have recurred following definitive therapy with any combination of surgery, radiation, and/or chemotherapy.
* All patients must have undergone salvage surgery in an attempt to excise all recurrent disease.
* Salvage radiation therapy must not be an option available to the patient.
* Patients must have high risk features such extra nodal invasion, positive margins, perineural invasion or vascular embolism.

Exclusion Criteria:

* Patients with macroscopic residual disease
* Patient is eligible for radiation therapy.
* Performance status more than 2.
* Contraindications for immunotherapy, autoimmune disease, allergy to medication, steroid use at baseline.
* Patients with other previous cancers excluding CIN, DCIS, non-melanoma skin cancers
* Patients previously treated with immunotherapy <12months prior
* Patients with synchronous cancers "not included in the inclusion criteria"

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Rate of recurrence at 1 year, will be measured by RECIST 1.1 as the primary measure for assessment of tumor, date of disease progression, and as a basis for all protocol guidelines related to disease status (e.g., discontinuation of study treatment). | 1 year
  Primary objective

SECONDARY OUTCOMES:
Determine the feasibility of immunotherapy for head and neck cancer following salvage surgery to produce preliminary data for 15 patients regarding efficacy. All side effects and symptoms will be assessed by CTCAE v5.0. | 1 year
  Study endpoint
Rate of completion of all planned therapy. All drug related toxicities will be graded by CTCAE v5.0. | through study completion, an average of 1 year
  Study endpoint
Toxicity rates measured by laboratory assessments and all adverse events and serious adverse events will be assessed by CTCAE v5.0. | through study completion, an average of 1 year
  Study endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Haythem Ali, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
This study is to obtain pilot data. The data may be shared with other researchers. Participants will sign a research HIPAA authorization to release their data. All participants will be assigned a study specific ID number.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after the study has completed enrollment and patient treatment. The data will be available indefinitely unless specified.
Access Criteria: Access will be limited to collaborators within and beyond Henry Ford Health System.